CLINICAL TRIAL: NCT01356277
Title: TAKE-IT: Teen Adherence in Kidney Transplant Effectiveness of Intervention Trial
Brief Title: Intervention to Improve Adherence in Teen Kidney Transplant
Acronym: TAKE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); Seattle Children's Hospital (Other); Washington University School of Medicine (Other); British Columbia Children's Hospital (Other); The Hospital for Sick Children (Other); St. Justine's Hospital (Other); Temple University (Other)
Responsible Party: Principal Investigator, Beth Foster, Associate Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01DK092977-01 (NIH)
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Kidney Transplantation; Medication Adherence
Keywords: renal; allograft; immunosuppressive; immunosuppression; adherence; medication; compliance
MeSH Terms: conditions — Medication Adherence; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-component Intervention (Experimental): Multi-component Intervention consisting of:
  * Adherence Support Team (patient, parent, Coach)
  * standardized education on immunosuppressive medications
  * identification of adherence barriers
  * Electronic adherence monitoring with feedback of past 3 months of electronic monitoring data at 3-month intervals
  * 'Action-Focused Problem-Solving' to address barriers selected as most important by the patient
  * text message, email, or visual cue dose reminders
  Interventions: Behavioral: Action-focused problem-solving; Device: Electronic pillbox monitoring, dose reminders, and feedback
- Attention control (No Intervention): Control group study visits were conducted at the same intervals as intervention visits and consisted of the Coach engaging in active listening and providing non-specific support only. Adherence was NOT discussed with control participants.

INTERVENTIONS:
Behavioral: Action-focused problem-solving — * Adherence Support Team (patient, parent, Coach)
  * standardized education on immunosuppressive medications
  * identification of adherence barriers
  * 'Action-Focused Problem-Solving' to address barriers selected as most important by the patient
  Arms: Multi-component Intervention
Device: Electronic pillbox monitoring, dose reminders, and feedback — * Electronic adherence monitoring with feedback of past 3 months of electronic monitoring data at 3-month intervals
  * text message, email, or visual cue dose reminders
  Other Names: Medminder Systems; Maya; US Patent Number 5710551; Vaica Medical; SimpleMed medication reminder and dispenser
  Arms: Multi-component Intervention

SUMMARY:
The broad aim of the proposed study is to improve medication adherence in adolescent kidney transplant recipients. The investigators hypothesize that a multi-component intervention will improve medication adherence in the adolescent kidney transplant population. The specific aims are to determine, in a randomized clinical trial, the efficacy of a structured, multi-component intervention in improving adherence to anti-rejection medications and graft outcomes, and to identify characteristics of healthcare systems that are independently associated with adherence.

DETAILED DESCRIPTION:
Young kidney transplant recipients at 8 pediatric transplant centers in the United States and Canada will be invited to participate. Participants will be randomly assigned to either the control or intervention group. Adherence will be measured in all participants using an electronic medication monitoring multi-dose pillbox. Enrolment will be followed by a 3-month run-in period, during which group allocation will be concealed and no intervention administered. At the 3-month visit, participants assigned to the intervention group will form an Adherence Support Team including the participant, one or both parents, and a study facilitator who is not a member of the treating team. At the same visit the facilitator will provide standardized adherence education, and will initiate a novel 20-30 min. behavioural intervention, which combines problem-solving skills with implementation intentions (concrete action plans in which an individual specifies, in an if-then contingency format, when, where and how he or she will perform a behaviour, with the goal of developing habits). This intervention will focus on addressing adherence barriers identified using the validated Medication Barriers Survey 3 and selected by the participant as important to him or her. Subsequent study visits, at 3-month intervals, will include a briefer versions of the educational component, and review and updating of implementation intentions. In addition, the electronic pillbox will be configured to provide alarm, phone, or text message dose reminders to participants in the intervention group throughout the intervention interval. Control participants will also meet with the facilitator at 3-month intervals, but will simply discuss general health and life issues; they will not receive dose reminders. In between visits, the facilitator will maintain monthly contact with all participants via short phone or text-message check-ins to troubleshoot issues with the electronic pillbox. The primary outcome will be 'taking adherence' - the proportion of prescribed doses that were consumed. Appropriate timing of doses will also be evaluated, as will variability in medication levels (reflecting consistency of medication consumption), and graft outcomes. Level of adherence, patterns of change in adherence, and graft outcomes will be compared between intervention and control groups. Secondary observational analyses of collected study data will identify healthcare systems factors independently associated with adherence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 11 - 24 years
* At least 3 months post kidney transplant

Exclusion Criteria:

* Significant neurocognitive disabilities limiting the subject's ability to understand and participate on their own
* Unable to communicate in English or French (Montreal site)
* Unable to communicate in English (all other sites)

Ages: 11 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2012-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany J Foster, MD, MSCE, Principal Investigator — Montreal Children's Hospital of the MUHC; Susan L Furth, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (8):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Canada (4):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - University of Toronto Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - St. Justine's Hospital, Montreal, Quebec

REFERENCES:
- [Background] Foster BJ, Pai A, Zhao H, Furth S; TAKE-IT Study Group. The TAKE-IT study: aims, design, and methods. BMC Nephrol. 2014 Aug 30;15:139. doi: 10.1186/1471-2369-15-139. PMID 25176317
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Boucquemont J, Pai ALH, Dharnidharka VR, Hebert D, Zelikovsky N, Amaral S, Furth SL, Foster BJ. Association between day of the week and medication adherence among adolescent and young adult kidney transplant recipients. Am J Transplant. 2020 Jan;20(1):274-281. doi: 10.1111/ajt.15590. Epub 2019 Oct 12. PMID 31507087
- [Derived] Boucquemont J, Pai ALH, Dharnidharka VR, Hebert D, Furth SL, Foster BJ. Gender Differences in Medication Adherence Among Adolescent and Young Adult Kidney Transplant Recipients. Transplantation. 2019 Apr;103(4):798-806. doi: 10.1097/TP.0000000000002359. PMID 29994983
- [Derived] Foster BJ, Pai ALH, Zelikovsky N, Amaral S, Bell L, Dharnidharka VR, Hebert D, Holly C, Knauper B, Matsell D, Phan V, Rogers R, Smith JM, Zhao H, Furth SL. A Randomized Trial of a Multicomponent Intervention to Promote Medication Adherence: The Teen Adherence in Kidney Transplant Effectiveness of Intervention Trial (TAKE-IT). Am J Kidney Dis. 2018 Jul;72(1):30-41. doi: 10.1053/j.ajkd.2017.12.012. Epub 2018 Mar 27. PMID 29602631

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient withdrew after completing the enrollment visit, but before randomization.
Groups:
- Behavioral Intervention: Participants in the intervention group will form an Adherence Support Team (AST), receive standardized adherence education, and complete behavioral intervention at 3-month intervals. In between visits, the study facilitator will maintain monthly contact with participants via short phone or text-message check-ins. The electronic pillbox will collect adherence data and will be configured to provide visual cue or text message dose reminders to participants in the intervention group. Participants in the intervention group will be fed back their electronic adherence data at each study visit.
  Action-focused problem-solving: An Adherence Support Team (AST), consisting of the patient, one or both parents (or primary caregiver), and the study facilitator, will be formed for each participant in the intervention arm. "Action-focused problem-solving" is informed by two complementary behavioral approaches: problem-solving and implementation intentions.
  Implementation intentions are concrete
- Attention Control: Control participants will receive an electronic pillbox to measure medication adherence. They will meet with the study facilitator at 3-month intervals to discuss general health and life issues. The dose reminder functions of the electronic pillbox will not be enabled.
Period: Run-in
Arm/Group | Behavioral Intervention | Attention Control
Started (Run-in) | 81 | 88
Completed (run-in) | 76 | 88
Not Completed | 5 | 0
Period: Intervention Interval
Arm/Group | Behavioral Intervention | Attention Control
Started | 76 | 88
Completed | 66 | 81
Not Completed | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Behavioral Intervention: Participants in the intervention group form an Adherence Support Team (AST), receive standardized adherence education, and complete behavioral intervention at 3-month intervals. In between visits, the study facilitator will maintain monthly contact with participants via short phone or text-message check-ins. The electronic pillbox will collect adherence data and will be configured to provide visual cue or text message dose reminders to participants in the intervention group. Participants in the intervention group will be fed back their electronic adherence data at each study visit.
  Action-focused problem-solving: An Adherence Support Team (AST), consisting of the patient, one or both parents (or primary caregiver), and the study facilitator, will be formed for each participant in the intervention arm. "Action-focused problem-solving" is informed by two complementary behavioral approaches: problem-solving and implementation intentions.
  Implementation intentions are concrete
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention | Attention Control | Total
Number analyzed (Participants) | 81 | 88 | 169
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15.5 [13.2 to 17.4] | 15.8 [13.3 to 17.4] | 15.8 [13.2 to 17.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 46 | 54 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 72 | 83 | 155
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 57 | 57 | 114
  Race: Black | 9 | 11 | 20
  Race: Asian | 4 | 7 | 11
  Race: Other | 11 | 13 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 27 | 32 | 59
  United States | 54 | 56 | 110
medication insurer [Count of Participants; unit: Participants]
  U.S. Public | 26 | 20 | 46
  Private | 28 | 36 | 64
  Canada provincial | 27 | 32 | 59
household income [Count of Participants; unit: Participants]
  < $25,000 | 19 | 10 | 29
  $25,000- $50,000 | 17 | 20 | 37
  $51,000- $75,000 | 17 | 22 | 39
  $76,000- $100,000 | 6 | 9 | 15
  >$100,000 | 12 | 16 | 28
  prefer not to answer | 5 | 2 | 7
  unknown | 5 | 9 | 14
median years post-transplant [Median (Inter-Quartile Range); unit: years] | 3.7 [0.7 to 7.9] | 3.0 [0.8 to 7.2] | 3.1 [0.7 to 7.5]
donor source [Count of Participants; unit: Participants]
  Living | 37 | 51 | 88
  Deceased | 44 | 37 | 81
median total lifetime duration of dialysis [Median (Inter-Quartile Range); unit: Months] | 10.0 [0.1 to 19.0] | 5.0 [0 to 12.0] | 6.0 [0.0 to 15.0]
primary disease [Count of Participants; unit: Participants]
  Congenital anomalies of the kidneys/ urinary tract | 29 | 41 | 70
  glomerulonephritis | 9 | 5 | 14
  Focal segmental glomerulosclerosis | 14 | 6 | 20
  other | 29 | 36 | 65
number of past acute rejections [Count of Participants; unit: Participants]
  0 | 59 | 76 | 135
  1 | 16 | 8 | 24
  2 or more | 6 | 4 | 10
number of comorbidities [Count of Participants; unit: Participants]
  0 | 41 | 43 | 84
  at least 1 | 40 | 45 | 85
number of doses of immunosuppressives per day [Median (Inter-Quartile Range); unit: number of doses per day] | 7 [5 to 9] | 7 [5 to 9] | 7 [5 to 9]
pre-intervention taking adherence [Number; unit: % days with 100% taking adherence] | 72.8 | 74.7 | 73.8
Total Adolescent Medication Barriers scale score [Mean (Standard Deviation); unit: units on a scale] — A higher Adolescent medication Barriers Scale (AMBS) represents a greater burden of barriers. The possible range for total score is 17-85.
  units on a scale | 37.5 (11.2) | 38.1 (9.8) | 37.7 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Taking Adherence
Description: Daily "taking adherence", defined as the percentage of prescribed doses taken each day (as measured by electronic monitoring). The daily taking adherence score could take a value of 0%, 50%, or 100% for patients on twice daily dosing, and 0% or 100% for patients on once daily dosing. Each patient had a taking adherence score for every day of observation (repeated measures). On days that the pillbox was not in use due to technical problems or participant non-use (due to travel etc), no score was given.
  To summarize adherence for each arm, we calculated the total percentage of days of observation for which there was 100% taking adherence. The denominator for this calculation was the the total number of days of observation of each participant, summed across all participants; the numerator was the total number of days of observation of each participant for which taking adherence was 100%, summed across all participants.
Time Frame: 12 months
Population: We used unadjusted ordinal logistic regression with generalized estimating equations to account for repeated measures (i.e. score on each day) to compare taking and timing adherence between the intervention and control groups during the intervention interval. An additional 'as-treated' analysis was also conducted. All available data were included.
Measure: Number; unit: % of days with 100% taking adherence
Groups:
- Behavioral Intervention: The patient, parent and Coach formed an Adherence Support Team. The Coach delivered standardized education on immunosuppressive medications, identified adherence barriers using the AMBS/PMBS and the last 3 months of electronic monitoring data and then used 'Action-Focused Problem-Solving' to address barriers selected as most important by the patient.
  Action-focused problem-solving involved brainstorming possible solutions to a barrier, rating the potential solutions, and selecting one solution to implement following the session. The solution was concrete and took the form of an "If/when…then…" statement. Intervention participants could choose to receive text message, email, or visual cue dose reminders. At subsequent sessions the Coach, patient, and parent jointly reviewed the electronic adherence monitoring data from the prior 3 mo to identify adherence patterns and guide the development and revision of action plans.
Arm/Group | Behavioral Intervention | Attention Control
Number analyzed (Participants) | 64 | 74
% of days with 100% taking adherence | 78 | 68
Statistical Analysis 1: Comparison: Behavioral Intervention vs Attention Control; We estimated a sample size of 75 participants per group to have 85% power to detect a 20% difference in taking adherence between groups, using 2-sided tests and setting alpha at 0.05, assuming a common standard deviation of 40%. Targeted enrollment of 176 participants accounted for 15% drop-out. Only participants with electronic pillbox data could be included. For participants who withdrew or stopped using the pillbox, all available pillbox data were included; Test type: Superiority; p = 0.006, Regression, Logistic; Unadjusted, ordinal logistic regression; Odds Ratio (OR) = 1.66, 95% CI 2-sided [1.15 to 2.39] — An odds ratio greater than 1.0 indicates higher adherence in Intervention participants compared with controls

2. Primary Outcome: Timing Adherence
Description: Daily "timing adherence", defined as the percentage of doses taken within 1 hour before to 2 hours after the prescribed dosing time each day (as measured by electronic monitoring). The daily timing adherence score could take a value of 0%, 50%, or 100% for patients on twice daily dosing, and 0% or 100% for patients on once daily dosing. Each patient had a timing adherence score for every day of observation (repeated measures). On days that the pillbox was not in use due to technical problems or participant non-use (due to travel etc), no score was given.
  To summarize timing adherence for each arm, we calculated the total percentage of days of observation for which there was 100% timing adherence. The denominator for this calculation was the the total number of days of observation of each participant, summed across all participants; the numerator was the total number of days of observation of each participant for which timing adherence was 100%, summed across all participants.
Time Frame: 12 months
Population: We used unadjusted ordinal logistic regression with generalized estimating equations to account for repeated measures (i.e. score on each day) to compare timing adherence between the intervention and control groups during the intervention interval. An additional 'as-treated' analysis was also conducted. All available data were included.
Measure: Number; unit: % of days with 100% timing adherence
Arm/Group | Behavioral Intervention | Attention Control
Number analyzed (Participants) | 64 | 74
% of days with 100% timing adherence | 73 | 61
Statistical Analysis 1: Comparison: Behavioral Intervention vs Attention Control; Test type: Superiority; p = 0.003, Regression, Logistic; Unadjusted ordinal logistic regression; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.21 to 2.50] — An odds ratio greater than 1.0 indicates higher adherence in Intervention participants compared with controls

3. Secondary Outcome: Standard Deviation (SD) of Tacrolimus Trough Levels
Description: The SD of all tacrolimus trough levels done for clinical care (except during hospitalizations or illnesses) were calculated for participants with >=3 tacrolimus levels.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: standard deviation units
Groups:
- Behavioral Intervention: Participants met with the coach at 3-month intervals. At each visit they had the opportunity to revise their Action plan or generate a new one. Action plans were concrete plans to address an adherence barrier that took the form "When... then..."
- Standard Care: Participants in the control group met with the coach at 3-month intervals but did not discuss adherence. They received general social support.
Arm/Group | Behavioral Intervention | Standard Care
Number analyzed (Participants) | 58 | 63
standard deviation units | 1.6 [0.9 to 2.5] | 1.4 [0.9 to 2.1]
Statistical Analysis 1: Comparison: Behavioral Intervention vs Standard Care; Null hypothesis was that there was no difference in the SD of tacrolimus trough levels between intervention and control; Test type: Superiority; p = 0.49, Wilcoxon ranksum

4. Secondary Outcome: Self-reported Taking Adherence
Description: Self-reported taking adherence, assessed using the Medical Adherence Measure- Medication Module (MAM-MM), was scored as the proportion of doses taken in the previous week. MAM-MM scores for each patient were summarized as the mean of the four scores post-intervention.
Time Frame: 12 months
Population: included all those who participated during the intervention interval
Measure: Mean (Standard Deviation); unit: percentage of prescribed doses taken
Arm/Group | Behavioral Intervention | Standard Care
Number analyzed (Participants) | 76 | 88
percentage of prescribed doses taken | 98.3 (4.5) | 97.1 (6.0)
Statistical Analysis 1: Comparison: Behavioral Intervention vs Standard Care; Test type: Superiority; p = 0.15, t-test, 2 sided

5. Secondary Outcome: Self-reported Timing Adherence
Description: Self-reported timing adherence, assessed using the Medical Adherence Measure- Medication Module (MAM-MM), was scored as the proportion of doses taken up to 2 hours after the prescribed time in the previous week. MAM-MM scores for each patient were summarized as the mean of the four scores post-intervention.
Time Frame: 12 months
Population: included all those who participated during the intervention interval
Measure: Mean (Standard Deviation); unit: percentage of doses taken on time
Arm/Group | Behavioral Intervention | Standard Care
Number analyzed (Participants) | 76 | 88
percentage of doses taken on time | 95.0 (7.9) | 92.9 (9.3)
Statistical Analysis 1: Comparison: Behavioral Intervention vs Standard Care; Test type: Superiority; p = 0.15, t-test, 2 sided

6. Secondary Outcome: Acute Rejection Rate
Description: The acute rejection rate, measured as rejections per 100 person-years of observation.
Time Frame: 12 months
Population: included all those who participated during the intervention interval
Measure: Number; unit: events per 100 person-years
Arm/Group | Behavioral Intervention | Standard Care
Number analyzed (Participants) | 76 | 88
events per 100 person-years | 1.06 | 1.69
Statistical Analysis 1: Comparison: Behavioral Intervention vs Standard Care; Rates were compared between intervention and control groups using Chi square; Test type: Superiority; p = 0.26, Chi-squared

7. Secondary Outcome: Annualized Change in Estimated Glomerular Filtration Rate (eGFR)
Description: Change in estimated glomerular filtration rate, estimated using the Schwartz equation for those < 18 y. and the CKD-EPI equation for those 18y and older, standardized to a 12-month period.
Time Frame: 12 months
Population: included all those with eGFR data available
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73m^2
Arm/Group | Behavioral Intervention | Standard Care
Number analyzed (Participants) | 66 | 81
ml/min/1.73m^2 | -2.3 [-10.6 to 2.3] | -3.3 [-7.7 to 3.7]
Statistical Analysis 1: Comparison: Behavioral Intervention vs Standard Care; Test type: Superiority; p = .45, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Description: The standard definitions were used.
Groups:
- Multi-component Intervention: * Adherence Support Team (patient, parent, Coach)
  * standardized education on immunosuppressive medications
  * identification of adherence barriers
  * Electronic adherence monitoring with feedback of past 3 months of electronic monitoring data at 3-month intervals
  * 'Action-Focused Problem-Solving' to address barriers selected as most important by the patient
  * text message, email, or visual cue dose reminders
- Attention Control: * Electronic adherence monitoring
  * meetings with Coach at 3 month intervals
Arm/Group | Multi-component Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/88
Serious Adverse Events (participants affected / at risk) | 24/76 | 30/88
Other Adverse Events (participants affected / at risk) | 42/76 | 52/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-component Intervention (N=76) | Attention Control (N=88)
Hospitalizations (General disorders) | 24 (42) | 29 (54)
PTLD (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-component Intervention (N=76) | Attention Control (N=88)
acute rejection (Renal and urinary disorders) | 8 (9) | 10 (17)
CMV infection (Infections and infestations) | 4 (5) | 0 (0)
influenza infection (Infections and infestations) | 3 (3) | 5 (5)
other infection (Infections and infestations) | 14 (20) | 21 (31)
vomiting/diarrhea (Gastrointestinal disorders) | 4 (5) | 3 (3)
surgery/procedure (Surgical and medical procedures) | 5 (7) | 6 (6)
Abdominal pain (General disorders) | 4 (5) | 7 (8)

LIMITATIONS AND CAVEATS:
Patients who withdrew or ceased to use the pillbox may introduce bias if they represented patients who were more or less adherent than those who continued to use the pillbox.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No